CLINICAL TRIAL: NCT02290184
Title: Pilipino Americans Go4Health Weight Loss Program to Prevent Heart Disease
Brief Title: PilAm Go4Health Weight Loss Program to Prevent Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Melinda Bender, Assistant Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14-14158; 14CRP19560008 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2014-11-08; First posted 2014-11-13 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Type2 Diabetes
Keywords: Type 2 diabetes; cardiovascular disease prevention; weight loss lifestyle intervention; physical activity; diet; Filipinos
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: statistician has been masked from any subjects' personal and confidential information
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention - PilAm Go4Health Program (Experimental): In the first 3 months this groups will start with the PilAm Go4Health Weight-loss Program lifestyle intervention. After 3 months this group will transition to a 3-month maintenance phase where they will continue to maintain the physical activity and healthy eating behaviors learned in the PilAm Go4Health Weight-loss Program lifestyle intervention and will complete the study for a total of 6 months.
  Interventions: Behavioral: PilAm Go4Health Weight-loss Program
- Active control - pedometer only (Active Comparator): In the first 3 months this groups will start with a pedometer only. After 3 months, this group will transition to receive the PilAm Go4Health Weight-loss Program lifestyle intervention for the next 3 month and will complete the study for a total of 6 months
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: PilAm Go4Health Weight-loss Program — This is a 3-month lifestyle intervention program promoting weight loss through physical activity and health diet using a mobile health application (app), pedometer to track daily step-counts, and social networking (in-person and virtual social networking through Facebook) to reduce risks for metabolic syndrome in Filipino Americans with type 2 diabetes on metformin. Subjects will be asked: 1) to use a mobile app diary every day to input their weight, and calories (food and drink intake) and 2) wear a pedometer everyday to monitor their physical activity (step-counts).
  Other Names: PilAm Go4Health Program
  Arms: Intervention - PilAm Go4Health Program
Behavioral: Active Control — This is a 3-month active control using a pedometer only without any education related to wt loss, physical activity, health eating, or tracking healthy behaviors
  Other Names: pedometer only
  Arms: Active control - pedometer only

SUMMARY:
This is a pilot randomized controlled trial intervention to improve lifestyle behaviors (physical activity and health diet) for Filipino Americans with type 2 diabetes on metformin. If the PilAm Go4Health intervention demonstrates potential efficacy, it may identify effective intervention strategies to significantly reduce risks for heart disease risks (i.e., metabolic syndrome) in Filipino Americans.

DETAILED DESCRIPTION:
Filipino Americans are the second largest Asian population and fastest growing racial group in the United States. They have one of the highest rates of insulin resistance (type 2 diabetes = T2DM) and central obesity (fat distributions primarily in the abdominal region). T2DM and central obesity are two of five major risk factors for metabolic syndrome that lead to cardiovascular disease and stroke. Key factors contributing to obesity and T2DM in Filipinos are their physical inactivity, and a diet high in fat and soda intake. However, there are very few research studies on improving health behaviors to reduce risks for metabolic syndrome in Filipino Americans. To help reduce the risk of developing metabolic syndrome in overweight/obese Filipino Americans with T2DM, the proposed project will test a culturally appropriate health behavior intervention program to reduce weight and waist circumference, through increasing physical activity, and lowering fat and sugar sweetened beverage intake. This intervention uses a mobile phone health app and social networking to encourage adherence to target health behaviors. The goals are to:

1. To assess feasibility and acceptability of the culturally appropriate PilAm Go4Health Weight Loss Program
2. To obtain preliminary estimates of the effect of the intervention on weight
3. To conduct post-program process evaluations too improve the intervention relevancy for the target population.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identified as Filipino
2. Age > 18 years
3. BMI for Asians > 23 kg/m2
4. Physician diagnosed T2DM diabetes confirmed by clinical data (e.g. documentation of fasting blood glucose >126 mg/dL or a positive oral glucose tolerance test (OGTT) > 200 mg/dl, HbA1c > 6.5%)
5. On metformin for T2DM

4) waist circumference: men > 40 inches, women > 35 inches 6) Physically inactive - most leisure time spent without much physical activity 7) No cognitive impairment per the Mini-Cog test 8) has a mobile smart phone (iPhone 4s or above, or android phone) 9) English speaking. Only one member per household allowed to enroll in the study.

Exclusion Criteria:

1. Uncontrolled T2DM
2. Glucose metabolism associated disease (Cushing's syndrome, Acromegaly, and Pheochromocytoma currently under treatment, chronic pancreatitis), 2) Thyroid disease - sub-optimally treated
3. Known medical conditions or other physical problems needing a special exercise program (e.g., prior myocardial infarction, history of angioplasty or angina, admission for hospital evaluation of chest pain, use of nitroglycerin for angina, chronic obstructive pulmonary disease, or uncontrolled hypertension)
4. Recent acute coronary syndrome, congestive heart failure
5. Currently participating in a lifestyle modification program
6. Planning a trip outside of the US during the 6-month study period
7. Known eating disorder
8. Planning a surgery in the next 7-months
9. Taking long-term antibiotics (including HIV-related agents), anti-tuberculosis agents (except isoniazid alone as prophylaxis), or prescription weight-loss drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda S Bender, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco / Daly City Communities, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated under this project will be administered in accordance with both University and NIH policies, including the NIH Data Sharing Policy and Implementation Guidance of March 5, 2003. That data set will be made available to qualified investigators within one year after completion of our investigators' data analyses and publication of papers presenting the results of those analyses.
  Requests will be reviewed and acted on by the PI or in consultation with a UCSF representative. After approval, the PI will prepare the requested dataset. This dataset will be carefully screened to make certain that all identifying information has been removed, including information that could be combined so as to identify an individual. Data will be provided in comma separated variables (CSV) text format rather than a proprietary format either on a CD or through a password-protected download from our website.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: That data set will be made available to qualified investigators within one year after completion of our investigators' data analyses and publication of papers presenting the results of those analyses.
Access Criteria: Data generated under this project will be administered in accordance with both University and NIH policies, including the NIH Data Sharing Policy and Implementation Guidance of March 5, 2003.Requests will be reviewed and acted on by the PI or in consultation with a University of California San Francisco (UCSF) representative. After approval, the PI will prepare the requested dataset. This dataset will be carefully screened to make certain that all identifying information has been removed, including information that could be combined so as to identify an individual. Data will be provided in comma separated variables (CSV) text format rather than a proprietary format either on a computer disk (CD) or through a password-protected download from our website.

REFERENCES:
- [Derived] Bender MS, Cooper BA, Park LG, Padash S, Arai S. A Feasible and Efficacious Mobile-Phone Based Lifestyle Intervention for Filipino Americans with Type 2 Diabetes: Randomized Controlled Trial. JMIR Diabetes. 2017 Dec 12;2(2):e30. doi: 10.2196/diabetes.8156. PMID 30291068
- [Derived] Bender MS, Santos GM, Villanueva C, Arai S. Development of a Mobile Phone-Based Weight Loss Lifestyle Intervention for Filipino Americans with Type 2 Diabetes: Protocol and Early Results From the PilAm Go4Health Randomized Controlled Trial. JMIR Res Protoc. 2016 Sep 8;5(3):e178. doi: 10.2196/resprot.5836. PMID 27608829

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All potential participants are invited to complete a pre-telephone screening. Those who pass the pre-telephone screening are potentially eligible to participate in the study and invited to attend a screening baseline visit where they are asked to complete a physical exam, serum blood tests, and a 2 week run-in period.
Pre-assignment Details: During the 2-week run-in, eligible participants are asked to wear Fitbit pedometer every day for 10 hours/day, take photos with their smart phone of each meal for 3 consecutive days, and email these photos to research study email.
  Those who pass the physical exam, serum lab test, and run-in period are then randomized to one of two study groups.
Groups:
- Intervention Group - Start With PilAm Go4Health Intervention: In the first 3 months intervention group start PilAm Go4Health lifestyle intervention. After initial 3-months participants will transition to a 3-month maintenance phase to maintain weight loss and learned lifestyle behaviors on their own. Group will complete the study at 6 months.
  PilAm Go4Health Weight-loss Program: This is a 3-month lifestyle intervention promoting weight loss through physical activity and health diet using a mobile health app, pedometer to track daily step-counts, and social networking (in-person and Facebook) to reduce risks for metabolic syndrome in Filipino Americans with type 2 diabetes on oral meds. Subjects will be asked: 1) log daily calorie/food intake and weekly wt. in mobile app diary and 2) wear a pedometer for 10hrs/day to monitor steps
- Active Wait-list Control Group - Start With Pedometer Only: In the first 3 months this groups will start with a pedometer only. After 3 months, this group will transition to receive the PilAm Go4Health Weight-loss Program lifestyle intervention for the next 3 month and will complete the study for a total of 6 months
  PilAm Go4Health Weight-loss Program: This is a 3-month lifestyle intervention program promoting weight loss through physical activity and health diet using a mobile health application (app), pedometer to track daily step-counts, and social networking (in-person and virtual social networking through Facebook) to reduce risks for metabolic syndrome in Filipino Americans with type 2 diabetes on metformin. Subjects will be asked: 1) to use a mobile app diary every day to input their weight, and calories (food and drink intake) and 2) wear a pedometer everyday to monitor their physical activity (step-counts).
Period: Overall Study
Arm/Group | Intervention Group - Start With PilAm Go4Health Intervention | Active Wait-list Control Group - Start With Pedometer Only
Started | 22 | 23
3-month Follow-up | 22 (Completed initial 3-month intervention and now transition to a 3-month maintenance phase) | 23 (Completed initial 3-month control period and transition to receive the 3-month intervention)
Completed | 22 (6-month follow-up visit - completed the 3-month maintenance phase and completed study) | 23 (6-month follow up visit - completed 3-month intervention and competed study)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Start With PilAm Go4Health Program: Baseline to 3-months this groups will start with the PilAm Go4Health Weight-loss Program lifestyle intervention. After 3 months this group will transition to a 3-month maintenance phase where they will continue to maintain the physical activity and healthy eating behaviors learned in the PilAm Go4Health Weight-loss Program lifestyle intervention and will complete the study for a total of 6 months.
  PilAm Go4Health Weight-loss Program: This is a 3-month lifestyle intervention program promoting weight loss through physical activity and health diet using a mobile health application (app), pedometer to track daily step-counts, and social networking (in-person and virtual social networking through Facebook) to reduce risks for metabolic syndrome in Filipino Americans with type 2 diabetes on metformin. Subjects will be asked: 1) to use a mobile app diary every day to input their weight, and calories (food and drink intake) and 2) wear a pedometer everyday to monitor physical activity
- Start With Pedometer Only: In the first 3 months this groups will start with a pedometer only. After 3 months, this group will transition to receive the PilAm Go4Health Weight-loss Program lifestyle intervention for the next 3 month and will complete the study for a total of 6 months
  PilAm Go4Health Weight-loss Program: This is a 3-month lifestyle intervention program promoting weight loss through physical activity and health diet using a mobile health application (app), pedometer to track daily step-counts, and social networking (in-person and virtual social networking through Facebook) to reduce risks for metabolic syndrome in Filipino Americans with type 2 diabetes on metformin. Subjects will be asked: 1) to use a mobile app diary every day to input their weight, and calories (food and drink intake) and 2) wear a pedometer everyday to monitor their physical activity (step-counts).
- Total: Total of all reporting groups
Arm/Group | Start With PilAm Go4Health Program | Start With Pedometer Only | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 23 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (9.8) | 57.7 (10.0) | 57.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 23 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 22 | 23 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Feasibility for Participant Enrollment and Retention
Description: Able to enroll at least 20 eligible participants per arm (measured by count), and retain at least 80% of enrolled participants in each arm
Time Frame: Baseline to 6-months
Population: Total number of enrolled participants in each arm who completed 6-month program divided by the total number of enrolled participants in each arm. Goal is to retain 80% of participants enrolled in each arm.
Measure: Number; unit: percentage of participants retained
Units Other Than Participants: participants
Groups:
- Intervention / PilAm Go4Health Program: In the first 3 months the Intervention group starts with the PilAm Go4Health Weight-loss Program lifestyle intervention. After 3 months the Intervention group transitions to a 3-month maintenance phase and continues physical activity and healthy eating behaviors learned in the PilAm Go4Health lifestyle intervention and then complete the study at the end of 6 months.
  PilAm Go4Health Weight-loss Program: This is a 3-month lifestyle intervention program promoting weight loss through physical activity and health diet using a mobile health application (app), pedometer to track daily step-counts, and social networking (in-person and virtual social networking through Facebook) to reduce risks for metabolic syndrome in Filipino Americans with type 2 diabetes on metformin. Subjects will be asked: 1) to use a mobile app diary every day to input their weight, and calories (food and drink intake) and 2) wear a pedometer everyday to monitor their physical activity (step-counts).
- Active Control - Pedometer Only: This group start the first 3-months with a pedometer only. After 3 months, this Active Control transitions to receive the PilAm Go4Health lifestyle intervention for the second 3 month and completes the study at the end of 6 months
  PilAm Go4Health Weight-loss Program: This is a 3-month lifestyle intervention program promoting weight loss through physical activity and health diet using a mobile health application (app), pedometer to track daily step-counts, and social networking (in-person and virtual social networking through Facebook) to reduce risks for metabolic syndrome in Filipino Americans with type 2 diabetes on metformin. Subjects will be asked: 1) to use a mobile app diary every day to input their weight, and calories (food and drink intake) and 2) wear a pedometer everyday to monitor their physical activity (step-counts).
Arm/Group | Intervention / PilAm Go4Health Program | Active Control - Pedometer Only
Number analyzed (Participants) | 22 | 23
percentage of participants retained | 22 | 23

2. Secondary Outcome: Weight Change in Kilograms
Description: weight change in kilograms over a 3 month period. Intervention group will have a significantly greater reduction in weight change compared to the active control from baseline to 3-months
Time Frame: Baseline to 3 months
Population: English-speaking Filipino Americans adults 18 years or older with overweight and Type 2 diabetes were randomized in a 1:1 ratio to either the intervention or active control group.
Measure: Mean (95% Confidence Interval); unit: kilogram
Arm/Group | Intervention Group - Start With PilAm Go4Health Intervention | Active Wait-list Control Group - Start With Pedometer Only
Number analyzed (Participants) | 22 | 23
kilogram | -2.1 [-2.9 to -1.4] | -.12 [-.72 to .59]
Statistical Analysis 1: Comparison: Intervention Group - Start With PilAm Go4Health Intervention vs Active Wait-list Control Group - Start With Pedometer Only; Hypothesis: the intervention group will have a significantly greater reduction in weight (kg) compared to the active control from baseline to 3-months; Test type: Superiority or Other — A multi-level regression was employed to test differences between the 2 arm's change trajectories of their estimated simple slopes. Bootstrapped full information maximum likelihood models were estimated to obtain nonparametric, bias-corrected confidence interval (CI); cross-level interaction = -2.0, .05% CI 2-sided [-3.0 to -1.1] — Multilevel regression analysis was used. The primary test of between-group change "effect" is also called the cross-level interaction between time and group. Simple slopes were also tested to determine if the change was significant within each group

3. Secondary Outcome: Percent Change in Weight (kg) From Baseline and 3 Months
Description: 100 x change in weight (kg) at 3 months divided by weight (kg) at baseline. Intervention group will have a significantly greater reduction in % weight change compared to the active control from baseline to 3-months.
Time Frame: Baseline to 3 months
Population: Filipino American adults 18 years or older with overweight and Type 2 diabetes were randomized in a 1:1 ratio to either the Intervention or the Active Control group.
Measure: Mean (95% Confidence Interval); unit: percent change
Groups:
- Intervention - PilAm Go4Health Program: Baseline to 3 months this groups will start with the PilAm Go4Health Weight-loss Program lifestyle intervention. After 3 months this group will transition to a 3-month maintenance phase where they will continue to maintain the physical activity and healthy eating behaviors learned in the PilAm Go4Health Weight-loss Program lifestyle intervention and will complete the study for a total of 6 months.
  PilAm Go4Health Weight-loss Program: This is a 3-month lifestyle intervention program promoting weight loss through physical activity and health diet using a mobile health application (app), pedometer to track daily step-counts, and social networking (in-person and virtual social networking through Facebook) to reduce risks for metabolic syndrome in Filipino Americans with type 2 diabetes on metformin. Subjects will be asked: 1) to use a mobile app diary every day to input their weight, and calories (food and drink intake) and 2) wear a pedometer everyday to monitor physical activity
- Active Control - Pedometer Only: In the first 3 months this groups will start with a pedometer only. After 3 months, this group will transition to receive the PilAm Go4Health Weight-loss Program lifestyle intervention for the next 3 month and will complete the study for a total of 6 months
  PilAm Go4Health Weight-loss Program: This is a 3-month lifestyle intervention program promoting weight loss through physical activity and health diet using a mobile health application (app), pedometer to track daily step-counts, and social networking (in-person and virtual social networking through Facebook) to reduce risks for metabolic syndrome in Filipino Americans with type 2 diabetes on metformin. Subjects will be asked: 1) to use a mobile app diary every day to input their weight, and calories (food and drink intake) and 2) wear a pedometer everyday to monitor their physical activity (step-counts).
Arm/Group | Intervention - PilAm Go4Health Program | Active Control - Pedometer Only
Number analyzed (Participants) | 22 | 23
percent change | -2.9 [-3.9 to -2.0] | -.28 [-1.0 to 0.56]
Statistical Analysis 1: Comparison: Intervention - PilAm Go4Health Program vs Active Control - Pedometer Only; Hypothesis: Intervention group will have a significantly greater reduction in % weight change compared to the active control from baseline to 3-months; Test type: Superiority — Multi-level regression was used to test differences between the 2 arm's change trajectories of their estimated simple slopes. Bootstrapped full information maximum likelihood models were estimated to obtain nonparametric, bias-corrected CI; cross-level interaction = -2.6, .05% CI 2-sided [-3.9 to -1.4] — Multilevel regression was used. The primary test of between group change "effect" is also called the cross-level interaction between time and group. Simple slopes were also tested to determine if the change was significant within each group

4. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference over time within groups
Time Frame: baseline to 3 months
Population: Multilevel regression used to analyze the within group change for waist circumference and cross-level interaction for between group change over time.
Measure: Mean (95% Confidence Interval); unit: centimeter
Groups:
- Start With PilAm Go4Health Program: Baseline to 3 months this groups will start with the PilAm Go4Health Weight-loss Program lifestyle intervention. At 3 months this group will begin a 3-month maintenance and will continue to maintain the physical activity and healthy eating behaviors learned in the PilAm Go4Health Weight-loss Program lifestyle intervention and will complete the study for a total of 6 months.
  PilAm Go4Health Weight-loss Program: This is a 3-month lifestyle intervention program promoting weight loss through physical activity and health diet using a mobile health application (app), pedometer to track daily step-counts, and social networking (in-person and virtual social networking through Facebook) to reduce risks for metabolic syndrome in Filipino Americans with type 2 diabetes on metformin. Subjects will be asked: 1) to use a mobile app diary every day to input their weight, and calories (food and drink intake) and 2) wear a pedometer everyday to monitor their physical activity (step-counts).
Arm/Group | Start With PilAm Go4Health Program | Start With Pedometer Only
Number analyzed (Participants) | 22 | 23
centimeter | -2.5 [-3.83 to -1.4] | -0.16 [-1.1 to 1.5]
Statistical Analysis 1: Comparison: Start With PilAm Go4Health Program vs Start With Pedometer Only; Hypothesis: Intervention group will have a significantly greater reduction in waist-circumference (cm) compared to the Active Control from baseline to 3-months; Test type: Superiority — A multi-level regression was used to test differences between the 2 arm's change trajectories of their estimated simple slopes. Bootstrapped full information maximum likelihood models were estimated to obtain nonparametric, bias-corrected CI; cross-level interaction = -2.7, 95% CI 2-sided [-4.5 to -.91] — Multilevel regression was used. The primary test of between -group change "effect" is also called the cross-level interaction between time and group. Simple slopes were also tested to determine if the change was significant within each group

ADVERSE EVENTS:
Time Frame: 13 months (Dec 2014 through Dec 2015)
Description: This study complied with the same clinicaltrials.gov definition for adverse event and/or serious adverse event. At each participant's schedule research office visit, an adverse event questionnaire was completed by the research staff to assess if any participant adverse events and/or serious adverse events had occurred since the previous research office visit.
Groups:
- Intervention - PilAm Go4Health Program: Baseline to 3 months this groups will start with the PilAm Go4Health Weight-loss Program lifestyle intervention. The intervention group will transition to a 3-month maintenance phase where they will continue to maintain the physical activity and healthy eating behaviors learned in the PilAm Go4Health Weight-loss Program lifestyle intervention and will complete the study for a total of 6 months.
  PilAm Go4Health Weight-loss Program: This is a 3-month lifestyle intervention program promoting weight loss through physical activity and health diet using a mobile health application (app), pedometer to track daily step-counts, and social networking (in-person and virtual social networking through Facebook) to reduce risks for metabolic syndrome in Filipino Americans with type 2 diabetes on metformin. Subjects will be asked: 1) to use a mobile app diary every day to input their weight, and calories (food and drink intake) and 2) wear a pedometer everyday to monitor their physical activity
Arm/Group | Intervention - PilAm Go4Health Program | Active Control - Pedometer Only
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23

LIMITATIONS AND CAVEATS:
Due to the study's small sample size and sample recruitment to one geographical region, study results cannot be generalized to other populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No